CLINICAL TRIAL: NCT00839696
Title: Total Xenoestrogen Body Burden in Relation to Mammographic Density, a Marker of Breast Cancer Risk
Brief Title: Total Xenoestrogen Body Burden in Relation to Mammographic Density, a Marker of Breast Cancer Rlisk
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CC07104; 2008-1013 (Other: Institutional Review Board); A538500 (Other: UW Madison); SMPH/POP HEALTH SCI (Other: UW Madison)
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2014-12

CONDITIONS: Breast Cancer Risk
Keywords: Breast; Estrogens; Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Xenoestrogen
Oversight: Data Monitoring Committee: No

SUMMARY:
Mammographic density is sensitive to estorgen exposure and constitutes a strong intermediate maker of breast cancer risk. We hypothesize that women with higher serum xenoestrogen levels will have greater mammographic density.

ELIGIBILITY:
Inclusion Criteria:

* 55-70 years of age, Post menopausal

Exclusion Criteria:

* If they have ever used hormone replacment therapy or have ever used Tamoxifen or Raloxifene, Diag. with breast cancer have had breast implants or have had a mastectomy/

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects recruited from screening mammography population
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Characterize the distribution of total xenoestrogen burden and identify important source of xenoestrogen exposure among a clinic-based sample of postmenopausal women. | 1 year

SECONDARY OUTCOMES:
Evaluate the association of total xenoestorgen exposure with mammographic density. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amy Trentham Dietz, PhD, Principal Investigator — Associate Professor- Population Health Sciences, UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin Hospital, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu